CLINICAL TRIAL: NCT03431246
Title: Persistance of Anti-HPV After a Single Dose of Gardasil and the Effect of a Dose of Gardasil-9 When Administered 3-8 Years Later
Brief Title: Immunogenicity of One Dose of Gardasil and One Dose of Gardasil-9
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Vladimir Gilca, Medical Epidemiologist, Laval University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CÉ: 2017-3036-21
Record Dates: First submitted 2018-01-26; First posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Human Papillomavirus Vaccines
MeSH Terms: interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Intervention Model Description: Single group exploratory study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gardasil and Gardasil-9 (Experimental)
  Interventions: Biological: Gardasil and Gardasil-9

INTERVENTIONS:
Biological: Gardasil and Gardasil-9 — All subjects will receive one dose of Gardasil-9. Blodd samples for serological testing will be collected just before and one month post Gardasil-9 administration.

SUMMARY:
This study will assess the immunogenicity of one dose of Gardasil and one dose of Gardasil-9

DETAILED DESCRIPTION:
This is a one group exploratory study.

The main objective of this study is to assess the persistance of anti-HPV after a single dose Gardasil and the effect of one dose of Gardasil-9 when administered 3-8 years later.

ELIGIBILITY:
Inclusion Criteria: Have received a single dose of Gardasil 3-8 years before recruitement.

-

Exclusion Criteria: Immunossupressed or blood coagulation problems

-

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Based on self-representation of gender identity
Enrollment: 32 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2016-11-05 (Actual); Study Completion 2016-12-05 (Actual)

PRIMARY OUTCOMES:
Anti-HPV seropositivity | One month post vaccine administration.
  Seropositivity to 9 HPV types included in Gardasil-9 vaccine will be assessed.

SECONDARY OUTCOMES:
HPV antibody titers | One month post vaccine administration
  Geometrical mean titers of antibodies to 9 HPV types included in Gardasil-9 vaccine will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Gaston DeSerres, MD, PhD, Study Chair — Quebec Public Health Institute
Locations (1):
- Laval University Research Hospital Center, Québec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guzun N, Ouakki M, Panicker G, Ionescu IG, Mayrand MH, Unger ER, Sauvageau C. Immune response after one dose of HPV vaccine among girls and boys and the impact of a second dose given after 3 or more years. Vaccine. 2025 Aug 30;62:127475. doi: 10.1016/j.vaccine.2025.127475. Epub 2025 Jul 14. PMID 40664165
- [Derived] Gilca V, Sauvageau C, Panicker G, De Serres G, Schiller J, Ouakki M, Unger ER. Long intervals between two doses of HPV vaccines and magnitude of the immune response: a post hoc analysis of two clinical trials. Hum Vaccin Immunother. 2019;15(7-8):1980-1985. doi: 10.1080/21645515.2019.1605278. Epub 2019 Jun 3. PMID 31017850